CLINICAL TRIAL: NCT02927457
Title: A Double-blind (Sponsor Unblinded) Study to Investigate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Clinical Effect of Repeat Dosing of GSK2646264 in Cutaneous Lupus Erythematosus Patients
Brief Title: Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Clinical Effect of GSK2646264 in Cutaneous Lupus Erythematosus Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 204860; 2016-000277-20 (EudraCT Number)
Record Dates: First submitted 2016-08-30; First posted 2016-10-07 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Lupus Erythematosus, Cutaneous
Keywords: Cutaneous Lupus Erythematosus-CLE; Spleen Tyrosine Kinase-SYK; Photoprovocation-PV; GSK2646264
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group A1- Skin Sites A/C/D (A/P/A) (Experimental): Skin areas A to E in group A are identified skin areas across the back of the subject. Subjects will be receiving GSK2646264 1% (A) for Area A- PV lesion, Placebo (P) for Area C- PV lesion and GSK2646264 1% for Area D- uninvolved skin once daily for 28 days according to randomisation. Skin areas B- PV lesion and E- uninvolved skin will not be assigned any treatment and will be used for the baseline biopsy.
  Interventions: Drug: GSK2646264 1%; Drug: Placebo
- Group A2- Skin Sites A/C/D (A/P/P) (Experimental): Skin areas A to E in group A are identified skin areas across the back of the subject. Subjects will be receiving GSK2646264 1% for Area A- PV lesion, Placebo for Area C- PV lesion and Placebo for Area D- uninvolved skin once daily for 28 days according to randomisation. Skin areas B- PV lesion and E- uninvolved skin will not be assigned any treatment and will be used for the baseline biopsy.
  Interventions: Drug: GSK2646264 1%; Drug: Placebo
- Group A3- Skin Sites A/C/D (P/A/A) (Experimental): Skin areas A to E in group A are identified skin areas across the back of the subject. Subjects will be receiving Placebo for Area A- PV lesion, GSK2646264 1% for Area C- PV lesion and GSK2646264 1% for Area D- uninvolved skin once daily for 28 days according to randomisation. Skin areas B- PV lesion and E- uninvolved skin will not be assigned any treatment and will be used for the baseline biopsy.
  Interventions: Drug: GSK2646264 1%; Drug: Placebo
- Group A4- Skin Sites A/C/D (P/A/P) (Experimental): Skin areas A to E in group A are identified skin areas across the back of the subject. Subjects will be receiving Placebo for Area A- PV lesion, GSK2646264 1% for Area C- PV lesion and Placebo for Area D- uninvolved skin once daily for 28 days according to randomisation. Skin areas B- PV lesion and E- uninvolved skin will not be assigned any treatment and will be used for the baseline biopsy.
  Interventions: Drug: GSK2646264 1%; Drug: Placebo
- Group B1- Skin Sites F/ G (A/P) (Experimental): In group B, two chosen lesions will be labeled F and G based on size (F >G). Subjects will be receiving GSK2646264 1% for lesion F and Placebo for lesion G once daily for 28 days according to randomisation. Skin area H- uninvolved skin will not be assigned any treatment and will be used for the baseline biopsy.
  Interventions: Drug: GSK2646264 1%; Drug: Placebo
- Group B2- Skin Sites F/ G (P/A) (Experimental): In group B, two chosen skin lesions will be labeled F and G based on size (F >G). Subjects will be receiving Placebo for lesion F and GSK2646264 1% for lesion G once daily for 28 days according to randomisation. Skin area H- uninvolved skin will not be assigned any treatment and will be used for the baseline biopsy.
  Interventions: Drug: GSK2646264 1%; Drug: Placebo

INTERVENTIONS:
Drug: GSK2646264 1% — A cream for topical application with a concentration of 1% GSK2646264.
Drug: Placebo — Subjects will receive matching Placebo topically.

SUMMARY:
This study is designed to examine safety, tolerability, pharmacokinetics, pharmacodynamics and clinical effect of repeat dosing of GSK2646264 in patients with subacute and chronic cutaneous lupus erythematosus (CLE) lesions and in acute CLE like lesions induced by photoprovocation (PV).

Current study is two group study. In Group A, Patients with fewer than two active lesions will be enrolled and exposed to photoprovocation (PV) for 3 consecutive days. Patients that develop PV lesions at any time during this period, as determined by the local investigative team, will receive 1% strength GSK2646264 on 1 lesion and placebo on 1 lesion daily and either 1% strength GSK2646264 or placebo on an area of uninvolved skin, for skin pharmacokinetic (PK) of study drug, for 28 days.

In Group B, Patients that have a minimum of 2 active existing CLE lesions as determined by the investigators will be enrolled into group B and have one lesion treated with 1% GSK2646264 and 1 lesion with placebo.

A completed patient will be defined as a subject who receives at least 25 days of study drug and completes the end of treatment biopsy (at day 28) and assessment. Thereafter patients will be followed for 28 days in Group A only or until complete resolution of induced PV lesions, as determined by the investigator.

ELIGIBILITY:
Inclusion Criteria

* Between 18 and 70 years of age inclusive, at the time of signing the informed consent.
* Subject values for the following parameters thyroid-stimulating hormone (TSH), free thyroxine (T4), and free triiodothyronine (T3) within the normal range.
* Subject has confirmed diagnosis of Lupus Erythematosus Tumidus (LET) (group A only), subacute or chronic CLE as determined by the investigators.
* Body weight >= 50 kg and body mass index (BMI) within the range 19.9 - 35 kilogram (kg)/meter square (m^2) (inclusive)
* Male OR Female.

Females: Non-reproductive potential defined as:

* Pre-menopausal females with one of the following: Documented tubal ligation, Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion , Hysterectomy, Documented Bilateral Oophorectomy
* Postmenopausal defined as 12 months of spontaneous amenorrhea. In questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 28 days prior to the first dose of study medication and until 12 days after the last dose of study medication and completion of the follow-up visit.

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.
* All subjects must be free from scarring or skin markings (e.g. tattoos or piercings) and open wounds on the defined areas of the body that cream will be applied onto or that will be exposed to PV, unless in the opinion of the investigator it will not compromise the subjects' safety and quality of data.
* Able to refrain from exposure to extended and direct sunlight during the study period, from screening until follow up, especially the area that is under treatment during the study.
* Able to refrain from using self-tanning products on the areas on which the study cream will be applied for the duration of the study from screening to follow-up.
* Able to refrain from shaving and waxing the areas on which the study cream will be applied during the duration of the study from screening to follow up.
* Patient stable on either no treatment or on :

  * Corticosteroids (=<7.5milligram [mg]/day prednisone or prednisone equivalent or less) for a minimum of 30 days prior to screening and through to Day 28.
  * and /or hydroxychloroquine (=<400mg daily dose) for a minimum of 60 days prior to the initial photoprovocation for group A or Randomisation Visit for group B through to day 28.
  * Topical steroids applied to the defined areas of the body that are not exposed to photoprovocation or study cream from screening to Day 28.
  * Topical calcineurin inhibitors and retinoids applied to the defined areas of the body that are not exposed to photoprovocation or study cream from screening to Day 28.

Exclusion Criteria

* ALT >2xupper limit of normal (ULN);
* Bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* QTcF > 450 millisecond (msec), or QTcF > 480 msec in subjects with Bundle Branch Block
* History of any past or present benign or malignant skin conditions and disease, unless in the opinion of the investigator it will not compromise the subjects safety and quality of data.
* Subjects with a history of Graves disease
* Subjects with a history of thyroid cancer.
* Unable to refrain from vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half lives (whichever is longer) prior to the screening visit until the completion of the follow-up assessments, unless in the opinion of the Investigator, in consultation with the GlaxoSmithKline (GSK) Medical Monitor if required, the medication will not interfere with the study procedures or compromise subject safety.
* Clinically significant abnormality in the hematological, clinical chemistry, or urinalysis screen, as judged by the investigator after discussion with the medical monitor.
* Subjects who start prohibited medications or therapies at any time during the study may be withdrawn from the study. Subjects who start prohibited medications or therapies may remain in the study only with the approval of the Medical Monitor and at the discretion of the Sponsor.
* The following medications and therapies are prohibited at any time during the study:

  * Use of other investigational agents (biologic or non-biologic; investigational applies to any drug not approved for sale in the country in which it is used).
  * Co-enrolment into another study of an investigational agent or non-drug therapy.
  * Use of biological agents (e.g., alemtuzumab [ATG], rituximab,) during the clinical study or within 12 months to first dose of study treatment.
  * Use of other immunosuppressive drugs commonly used in Systemic lupus erythematosus (SLE) including Azathioprine, Methotrexate, Mycophenolate, Cyclophosphamide within 3 months to first dose of study treatment.
* History of regular alcohol consumption within 3 months of the study defined as:

Alcohol will be allowed but limited to an average weekly intake of <21 units for males or <14 units for females).

* Direct exposure to ultraviolet (UV) light (e.g. sunbathing) to the testing areas within 2 weeks of study entry.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation (refer to the Investigator Brochure for a list of excipients).
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug screen.
* Where participation in the study would result in donation of blood or blood products in excess of 450 milliliter (ml) within 3 months.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than 4 investigational medicinal products within 12 months prior to the first dosing day.

Country Specific Exclusion criteria wording for Germany:

* Subjects that are employees of either GlaxoSmithKline (sponsor) or one of the study centres (investigators).
* Subjects who live in detention on court order or on regulatory action.
* Oral Prednisolone

  * Greater than 7.5 mg by mouth daily.
  * Any increase in dose from screening to Day 28
* Hydroxychloroquine

  * Greater than 400 mg oral daily.
  * Any increase in dose from screening to Day 28.
* Photosensitizing drugs within 5 half-lives prior to the photoprovocation visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Germany (5):
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Wuppertal, North Rhine-Westphalia
  - GSK Investigational Site, Berlin

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20789

REFERENCES:
- [Derived] Walker A, Erwig L, Foster K, Nevin K, Wenzel J, Worm M, Williams N, Ratia N, Hoang B, Schneider-Merck T, Gisbert S, Carnarius H, Dickson M. Safety, pharmacokinetics and pharmacodynamics of a topical SYK inhibitor in cutaneous lupus erythematosus: A double-blind Phase Ib study. Exp Dermatol. 2021 Nov;30(11):1686-1692. doi: 10.1111/exd.14253. Epub 2020 Dec 17. PMID 33336508

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a double blind (sponsor unblinded) Phase Ib two group [group A-photoprovocation (PV) lesions and group B-natural lesions] study to investigate repeat doses of GSK2646264 administered via topical delivery, on safety, pharmacodynamic effect and clinical efficacy in cutaneous lupus participants.
Pre-assignment Details: A total of 11 participants were enrolled in group B in this study. No participants were randomized in group A due to PV failure and feasibility. All participants in group B received both treatment interventions at the same time (on different skin sites), hence these participants were combined in the participant flow.
Groups:
- Group A-Participants With Photoprovocation Lesions: Participants who developed lesions following 3 consecutive days of photoprovocation were planned to be administered topical white to off-white GSK2646264 (1 percent [%] weight by weight [w/w]) to 1 lesion and placebo to 1 lesion (at the same time), once daily for 28 consecutive days. Either 1% w/w GSK2646264 or placebo was planned also to be administered to an area of uninvolved skin for 28 days.
- Group B-Participants With Natural Lesions: Participants with natural lesions were topically administered white to off-white aqueous cream of GSK2646264 (1% w/w) and placebo. The treatments were administered at the same time on different skin sites once daily for 28 days.
Period: Overall Study
Arm/Group | Group A-Participants With Photoprovocation Lesions | Group B-Participants With Natural Lesions
Started | 0 | 11
Completed | 0 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants received both treatment interventions at the same time (on different skin sites), hence, data for these participants were combined.
Groups:
- Group B- Participants With Natural Lesions: Participants with natural lesions were topically administered white to off-white aqueous cream of GSK2646264 (1% w/w) and placebo. The treatments were administered at the same time on different skin sites once daily for 28 days.
- Total: Total of all reporting groups
Arm/Group | Group A-Participants With Photoprovocation Lesions | Group B- Participants With Natural Lesions | Total
Number analyzed (Participants) | 0 | 11 | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] — All participants received both treatment interventions at the same time (on different skin sites), hence, data for these participants were combined.
  Years |  | 54.8 (10.44) | 54.8 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants] — All participants received both treatment interventions at the same time (on different skin sites), hence, data for these participants were combined.
  Participants
    Female | 0 | 9 | 9
    Male | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — All participants received both treatment interventions at the same time (on different skin sites), hence, data for these participants were combined.
  Participants
    Race: Black or African American | 0 | 1 | 1
    Race: White/Caucasian/European heritage | 0 | 10 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Emergent Chemistry Results by Potential Clinical Importance (PCI) Criteria
Description: Blood samples were collected to analyze the clinical chemistry parameters; albumin, alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (TB), calcium, glucose, potassium (Pot) and sodium. PCI ranges were albumin (low: <30 grams per liter), calcium (low: <2 millimoles per liter [mmol/L] and high: >2.75 mmol/L), glucose (low: <3 mmol/L and high: >9 mmol/L), Pot (low: <3 mmol/L and high: >5.5 mmol/L), sodium (low: <130 mmol/L and high: >150 mmol/L), ALT (high: >=2 times upper limit of normal [ULN] units per liter {U/L}), AST (high: >=2 times ULN U/L), ALP (high: >=2 times ULN U/L) and TB (high: >=1.5 times ULN micromoles per liter). Safety Population comprised of all participants who received at least one dose of study treatment. All participants received both treatment interventions at the same time (on different skin sites), hence data for these participants were combined.
Time Frame: Day 14, Day 28 and follow-up (up to Day 56)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles). Data was not collected for Group A as no participants were dosed.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A-Participants With Photoprovocation Lesions | Group B-Participants With Natural Lesions
Number analyzed (Participants) | 0 | 11
Participants
  Albumin, Day 14, To low, n=0,11 |  | 0
  Albumin, Day 14, To normal or no change, n=0,11 |  | 11
  Albumin, Day 28, To low, n=0,10: number analyzed (Participants) | 0 | 10
  Albumin, Day 28, To low, n=0,10 |  | 0
  Albumin, Day 28, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  Albumin, Day 28, To normal or no change, n=0,10 |  | 10
  Albumin, Follow-up, To low, n=0,11 |  | 0
  Albumin, Follow-up, To normal or no change, n=0,11 |  | 11
  ALP, Day 14, To normal or no change, n=0,11 |  | 11
  ALP, Day 14, To high, n=0,11 |  | 0
  ALP, Day 28, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  ALP, Day 28, To normal or no change, n=0,10 |  | 10
  ALP, Day 28, To high, n=0,10: number analyzed (Participants) | 0 | 10
  ALP, Day 28, To high, n=0,10 |  | 0
  ALP, Follow-up, To normal or no change, n=0,11 |  | 11
  ALP, Follow-up, To high, n=0,11 |  | 0
  ALT, Day 14, To normal or no change, n=0,11 |  | 11
  ALT, Day 14, To high, n=0,11 |  | 0
  ALT, Day 28, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  ALT, Day 28, To normal or no change, n=0,10 |  | 10
  ALT, Day 28, To high, n=0,10: number analyzed (Participants) | 0 | 10
  ALT, Day 28, To high, n=0,10 |  | 0
  ALT, Follow-up, To normal or no change, n=0,11 |  | 11
  ALT, Follow-up, To high, n=0,11 |  | 0
  AST, Day 14, To normal or no change, n=0,11 |  | 11
  AST, Day 14, To high, n=0,11 |  | 0
  AST, Day 28, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  AST, Day 28, To normal or no change, n=0,10 |  | 10
  AST, Day 28, To high, n=0,10: number analyzed (Participants) | 0 | 10
  AST, Day 28, To high, n=0,10 |  | 0
  AST, Follow-up, To normal or no change, n=0,11 |  | 11
  AST, Follow-up, To high, n=0,11 |  | 0
  TB, Day 14, To normal or no change, n=0,11 |  | 11
  TB, Day 14, To high, n=0,11 |  | 0
  TB, Day 28, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  TB, Day 28, To normal or no change, n=0,10 |  | 10
  TB, Day 28, To high, n=0,10: number analyzed (Participants) | 0 | 10
  TB, Day 28, To high, n=0,10 |  | 0
  TB, Follow-up, To normal or no change, n=0,11 |  | 11
  TB, Follow-up, To high, n=0,11 |  | 0
  Calcium, Day 14, To low, n=0,11 |  | 0
  Calcium, Day 14, To normal or no change, n=0,11 |  | 11
  Calcium, Day 14, To high, n=0,11 |  | 0
  Calcium, Day 28, To low, n=0,10: number analyzed (Participants) | 0 | 10
  Calcium, Day 28, To low, n=0,10 |  | 0
  Calcium, Day 28, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  Calcium, Day 28, To normal or no change, n=0,10 |  | 10
  Calcium, Day 28, To high, n=0,10: number analyzed (Participants) | 0 | 10
  Calcium, Day 28, To high, n=0,10 |  | 0
  Calcium, Follow-up, To low, n=0,11 |  | 0
  Calcium, Follow-up, To normal or no change, n=0,11 |  | 11
  Calcium, Follow-up, To high, n=0,11 |  | 0
  Glucose, Day 14, To low, n=0,11 |  | 0
  Glucose, Day 14, To normal or no change, n=0,11 |  | 11
  Glucose, Day 14, To high, n=0,11 |  | 0
  Glucose, Day 28, To low, n=0,10: number analyzed (Participants) | 0 | 10
  Glucose, Day 28, To low, n=0,10 |  | 0
  Glucose, Day 28, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  Glucose, Day 28, To normal or no change, n=0,10 |  | 10
  Glucose, Day 28, To high, n=0,10: number analyzed (Participants) | 0 | 10
  Glucose, Day 28, To high, n=0,10 |  | 0
  Glucose, Follow-up, To low, n=0,11 |  | 0
  Glucose, Follow-up, To normal or no change, n=0,11 |  | 11
  Glucose, Follow-up, To high, n=0,11 |  | 0
  Pot, Day 14, To low, n=0,11 |  | 0
  Pot, Day 14, To normal or no change, n=0,11 |  | 11
  Pot, Day 14, To high, n=0,11 |  | 0
  Pot, Day 28, To low, n=0,10: number analyzed (Participants) | 0 | 10
  Pot, Day 28, To low, n=0,10 |  | 0
  Pot, Day 28, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  Pot, Day 28, To normal or no change, n=0,10 |  | 10
  Pot, Day 28, To high, n=0,10: number analyzed (Participants) | 0 | 10
  Pot, Day 28, To high, n=0,10 |  | 0
  Pot, Follow-up, To low, n=0,11 |  | 0
  Pot, Follow-up, To normal or no change, n=0,11 |  | 11
  Pot, Follow-up, To high, n=0,11 |  | 0
  Sodium, Day 14, To low, n=0,11 |  | 0
  Sodium, Day 14, To normal or no change, n=0,11 |  | 11
  Sodium, Day 14, To high, n=0,11 |  | 0
  Sodium, Day 28, To low, n=0,10: number analyzed (Participants) | 0 | 10
  Sodium, Day 28, To low, n=0,10 |  | 0
  Sodium, Day 28, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  Sodium, Day 28, To normal or no change, n=0,10 |  | 10
  Sodium, Day 28, To high, n=0,10: number analyzed (Participants) | 0 | 10
  Sodium, Day 28, To high, n=0,10 |  | 0
  Sodium, Follow-up, To low, n=0,11 |  | 0
  Sodium, Follow-up, To normal or no change, n=0,11 |  | 11
  Sodium, Follow-up, To high, n=0,11 |  | 0

2. Primary Outcome: Number of Participants With Emergent Hematology Results by PCI Criteria
Description: PCI ranges were hematocrit [Hct] (high: >0.54 proportion of red blood cell [RBC] in blood), hemoglobin [Hb] (high: >180 grams per liter), RBC (low: <4.2x10^12 cells per liter and high: >5.9x10^12 cells per liter), lymphocytes [Lympho] (low: <0.8x10^9 cells per liter), monocytes [Mono] (low: <0.14x10^9 cells per liter and high: >1.3x10^9 cells per liter), neutrophils [Neutro] (low: <1.5x10^9 cells per liter), platelet count [PC] (low: <100x10^9 cells per liter and high: >550x10^9 cells per liter), eosinophils [Eos] (high: >0.55x10^9 cells per liter), basophils [Baso] (high: >0.22x10^9 cells per liter), white blood cell [WBC] (low: <3x10^9 cells per liter and high: >20x10^9 cells per liter). All participants received both treatment interventions at the same time (on different skin sites), hence data for these participants were combined.
Time Frame: Day 14, Day 28 and follow-up (up to Day 56)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A-Participants With Photoprovocation Lesions | Group B-Participants With Natural Lesions
Number analyzed (Participants) | 0 | 11
Participants
  Baso, Day 14, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  Baso, Day 14, To normal or no change, n=0,10 |  | 10
  Baso, Day 14, To high, n=0,10: number analyzed (Participants) | 0 | 10
  Baso, Day 14, To high, n=0,10 |  | 0
  Baso, Day 28, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  Baso, Day 28, To normal or no change, n=0,10 |  | 10
  Baso, Day 28, To high, n=0,10: number analyzed (Participants) | 0 | 10
  Baso, Day 28, To high, n=0,10 |  | 0
  Baso, Follow-up, To normal or no change, n=0,11 |  | 11
  Baso, Follow-up, To high, n=0,11 |  | 0
  Eos, Day 14, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  Eos, Day 14, To normal or no change, n=0,10 |  | 10
  Eos, Day 14, To high, n=0,10: number analyzed (Participants) | 0 | 10
  Eos, Day 14, To high, n=0,10 |  | 0
  Eos, Day 28, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  Eos, Day 28, To normal or no change, n=0,10 |  | 10
  Eos, Day 28, To high, n=0,10: number analyzed (Participants) | 0 | 10
  Eos, Day 28, To high, n=0,10 |  | 0
  Eos, Follow-up, To normal or no change, n=0,11 |  | 11
  Eos, Follow-up, To high n=0,11 |  | 0
  Hb, Day 14, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  Hb, Day 14, To normal or no change, n=0,10 |  | 10
  Hb, Day 14, To high, n=0,10: number analyzed (Participants) | 0 | 10
  Hb, Day 14, To high, n=0,10 |  | 0
  Hb, Day 28, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  Hb, Day 28, To normal or no change, n=0,10 |  | 10
  Hb, Day 28, To high, n=0,10: number analyzed (Participants) | 0 | 10
  Hb, Day 28, To high, n=0,10 |  | 0
  Hb, Follow-up, To normal or no change, n=0,11 |  | 11
  Hb, Follow-up, To high, n=0,11 |  | 0
  Hct, Day 14, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  Hct, Day 14, To normal or no change, n=0,10 |  | 10
  Hct, Day 14, To high, n=0,10: number analyzed (Participants) | 0 | 10
  Hct, Day 14, To high, n=0,10 |  | 0
  Hct, Day 28, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  Hct, Day 28, To normal or no change, n=0,10 |  | 10
  Hct, Day 28, To high, n=0,10: number analyzed (Participants) | 0 | 10
  Hct, Day 28, To high, n=0,10 |  | 0
  Hct, Follow-up, To normal or no change, n=0,11 |  | 11
  Hct, Follow-up, To high, n=0,11 |  | 0
  Lympho, Day 14, To low, n=0,10: number analyzed (Participants) | 0 | 10
  Lympho, Day 14, To low, n=0,10 |  | 0
  Lympho, Day 14, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  Lympho, Day 14, To normal or no change, n=0,10 |  | 10
  Lympho, Day 28, To low, n=0,10: number analyzed (Participants) | 0 | 10
  Lympho, Day 28, To low, n=0,10 |  | 0
  Lympho, Day 28, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  Lympho, Day 28, To normal or no change, n=0,10 |  | 10
  Lympho, Follow-up, To low, n=0,11 |  | 0
  Lympho, Follow-up, To normal or no change, n=0,11 |  | 11
  Mono, Day 14, To low, n=0,10: number analyzed (Participants) | 0 | 10
  Mono, Day 14, To low, n=0,10 |  | 0
  Mono, Day 14, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  Mono, Day 14, To normal or no change, n=0,10 |  | 10
  Mono, Day 14, To high, n=0,10: number analyzed (Participants) | 0 | 10
  Mono, Day 14, To high, n=0,10 |  | 0
  Mono, Day 28, To low, n=0,10: number analyzed (Participants) | 0 | 10
  Mono, Day 28, To low, n=0,10 |  | 1
  Mono, Day 28, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  Mono, Day 28, To normal or no change, n=0,10 |  | 9
  Mono, Day 28, To high, n=0,10: number analyzed (Participants) | 0 | 10
  Mono, Day 28, To high, n=0,10 |  | 0
  Mono, Follow-up, To low, n=0,11 |  | 0
  Mono, Follow-up, To normal or no change, n=0,11 |  | 11
  Mono, Follow-up, To high, n=0,11 |  | 0
  Neutro, Day 14, To low, n=0,10: number analyzed (Participants) | 0 | 10
  Neutro, Day 14, To low, n=0,10 |  | 1
  Neutro, Day 14, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  Neutro, Day 14, To normal or no change, n=0,10 |  | 9
  Neutro, Day 28, To low, n=0,10: number analyzed (Participants) | 0 | 10
  Neutro, Day 28, To low, n=0,10 |  | 0
  Neutro, Day 28, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  Neutro, Day 28, To normal or no change, n=0,10 |  | 10
  Neutro, Follow-up, To low, n=0,11 |  | 0
  Neutro, Follow-up, To normal or no change, n=0,11 |  | 11
  PC, Day 14, To low, n=0,10: number analyzed (Participants) | 0 | 10
  PC, Day 14, To low, n=0,10 |  | 0
  PC, Day 14, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  PC, Day 14, To normal or no change, n=0,10 |  | 10
  PC, Day 14, To high, n=0,10: number analyzed (Participants) | 0 | 10
  PC, Day 14, To high, n=0,10 |  | 0
  PC, Day 28, To low, n=0,10: number analyzed (Participants) | 0 | 10
  PC, Day 28, To low, n=0,10 |  | 0
  PC, Day 28, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  PC, Day 28, To normal or no change, n=0,10 |  | 10
  PC, Day 28, To high, n=0,10: number analyzed (Participants) | 0 | 10
  PC, Day 28, To high, n=0,10 |  | 0
  PC, Follow-up, To low, n=0,11 |  | 0
  PC, Follow-up, To normal or no change, n=0,11 |  | 11
  PC, Follow-up, To high, n=0,11 |  | 0
  RBC, Day 14, To low, n=0,10: number analyzed (Participants) | 0 | 10
  RBC, Day 14, To low, n=0,10 |  | 0
  RBC, Day 14, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  RBC, Day 14, To normal or no change, n=0,10 |  | 10
  RBC, Day 14, To high, n=0,10: number analyzed (Participants) | 0 | 10
  RBC, Day 14, To high, n=0,10 |  | 0
  RBC, Day 28, To low, n=0,10: number analyzed (Participants) | 0 | 10
  RBC, Day 28, To low, n=0,10 |  | 1
  RBC, Day 28, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  RBC, Day 28, To normal or no change, n=0,10 |  | 9
  RBC, Day 28, To high, n=0,10: number analyzed (Participants) | 0 | 10
  RBC, Day 28, To high, n=0,10 |  | 0
  RBC, Follow-up, To low, n=0,11 |  | 0
  RBC, Follow-up, To normal or no change, n=0,11 |  | 11
  RBC, Follow-up, To high, n=0,11 |  | 0
  WBC, Day 14, To low, n=0,10: number analyzed (Participants) | 0 | 10
  WBC, Day 14, To low, n=0,10 |  | 0
  WBC, Day 14, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  WBC, Day 14, To normal or no change, n=0,10 |  | 10
  WBC, Day 14, To high, n=0,10: number analyzed (Participants) | 0 | 10
  WBC, Day 14, To high, n=0,10 |  | 0
  WBC, Day 28, To low, n=0,10: number analyzed (Participants) | 0 | 10
  WBC, Day 28, To low, n=0,10 |  | 0
  WBC, Day 28, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  WBC, Day 28, To normal or no change, n=0,10 |  | 10
  WBC, Day 28, To high, n=0,10: number analyzed (Participants) | 0 | 10
  WBC, Day 28, To high, n=0,10 |  | 0
  WBC, Follow-up, To low, n=0,11 |  | 0
  WBC, Follow-up, To normal or no change, n=0,11 |  | 11
  WBC, Follow-up, To high, n=0,11 |  | 0

3. Primary Outcome: Change From Baseline in Urine Potential of Hydrogen (pH)
Description: Urine samples were collected to monitor the pH. pH is a measure of hydrogen ion concentration and is used to determine the acidity or alkalinity of urine. pH scale ranges from 0 to 14. A neutral pH is 7.0. The higher number indicates the more basic (alkaline) nature of urine and lower number indicates the more acidic urine. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. All participants received both treatment interventions at the same time (on different skin sites), hence data for these participants were combined.
Time Frame: Baseline (Day 1), Day 14, Day 28 and follow-up (up to Day 56)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Group A-Participants With Photoprovocation Lesions | Group B-Participants With Natural Lesions
Number analyzed (Participants) | 0 | 11
pH
  Day 14, n=0,10: number analyzed (Participants) | 0 | 10
  Day 14, n=0,10 |  | -0.10 (0.843)
  Day 28, n=0,10: number analyzed (Participants) | 0 | 10
  Day 28, n=0,10 |  | -0.35 (0.669)
  Follow-up, n=0,11 |  | -0.32 (0.783)

4. Primary Outcome: Change From Baseline in Urine Specific Gravity
Description: Urine samples were collected to monitor the specific gravity. Specific gravity is a measure of urine concentration and is measured using a chemical test. Specific gravity measurements provide a comparison of the amount of substances dissolved in urine as compared to pure water. If there were no solutes present, the specific gravity of urine would be 1.000 the same as pure water. Specific gravity between 1.002 and 1.035 could be considered as normal. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. All participants received both treatment interventions at the same time (on different skin sites), hence data for these participants were combined.
Time Frame: Baseline (Day 1), Day 14, Day 28 and follow-up (up to Day 56)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilogram per meter cube
Arm/Group | Group A-Participants With Photoprovocation Lesions | Group B-Participants With Natural Lesions
Number analyzed (Participants) | 0 | 11
kilogram per meter cube
  Day 14, n=0,10: number analyzed (Participants) | 0 | 10
  Day 14, n=0,10 |  | 0.0007 (0.00629)
  Day 28, n=0,10: number analyzed (Participants) | 0 | 10
  Day 28, n=0,10 |  | -0.0001 (0.00626)
  Follow-up, n=0,11 |  | 0.0003 (0.00746)

5. Primary Outcome: Number of Participants With Emergent Vital Sign Results by PCI Criteria
Description: Vital signs such as diastolic blood pressure (DBP), heart rate (HR) and systolic blood pressure (SBP) were measured in semi-supine position after 5 minutes rest for the participants. PCI ranges were SBP (lower: <85 millimeters of mercury [mmHg] and upper: >160 mmHg), DBP: (lower: <45 mmHg and upper: >100 mmHg) and HR (lower: <40 beats per minute [bpm] and upper: >110 bpm). All participants received both treatment interventions at the same time (on different skin sites), hence data for these participants were combined.
Time Frame: Day 14 and Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A-Participants With Photoprovocation Lesions | Group B-Participants With Natural Lesions
Number analyzed (Participants) | 0 | 11
Participants
  DBP, Day 14, To low, n=0,10: number analyzed (Participants) | 0 | 10
  DBP, Day 14, To low, n=0,10 |  | 0
  DBP, Day 14, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  DBP, Day 14, To normal or no change, n=0,10 |  | 10
  DBP, Day 14, To high, n=0,10: number analyzed (Participants) | 0 | 10
  DBP, Day 14, To high, n=0,10 |  | 0
  DBP, Day 28, To low, n=0,11 |  | 0
  DBP, Day 28, To normal or no change, n=0,11 |  | 11
  DBP, Day 28, To high, n=0,11 |  | 0
  HR, Day 14, To low, n=0,10: number analyzed (Participants) | 0 | 10
  HR, Day 14, To low, n=0,10 |  | 0
  HR, Day 14, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  HR, Day 14, To normal or no change, n=0,10 |  | 10
  HR, Day 14, To high, n=0,10: number analyzed (Participants) | 0 | 10
  HR, Day 14, To high, n=0,10 |  | 0
  HR, Day 28, To low, n=0,11 |  | 0
  HR, Day 28, To normal or no change, n=0,11 |  | 11
  HR, Day 28, To high, n=0,11 |  | 0
  SBP, Day 14, To low, n=0,10: number analyzed (Participants) | 0 | 10
  SBP, Day 14, To low, n=0,10 |  | 0
  SBP, Day 14, To normal or no change, n=0,10: number analyzed (Participants) | 0 | 10
  SBP, Day 14, To normal or no change, n=0,10 |  | 10
  SBP, Day 14, To high, n=0,10: number analyzed (Participants) | 0 | 10
  SBP, Day 14, To high, n=0,10 |  | 0
  SBP, Day 28, To low, n=0,11 |  | 0
  SBP, Day 28, To normal or no change, n=0,11 |  | 11
  SBP, Day 28, To high, n=0,11 |  | 0

6. Primary Outcome: Change From Baseline in Electrocardiogram (ECG); HR
Description: Triplicate 12-lead ECGs were obtained using an ECG machine that automatically calculated the heart rate. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. All participants received both treatment interventions at the same time (on different skin sites), hence data for these participants were combined.
Time Frame: Baseline (Day 1), Day 14 and follow-up (up to Day 56)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Group A-Participants With Photoprovocation Lesions | Group B-Participants With Natural Lesions
Number analyzed (Participants) | 0 | 11
bpm
  HR, Day 14, n=0,10: number analyzed (Participants) | 0 | 10
  HR, Day 14, n=0,10 |  | 1.633 (8.3702)
  HR, Follow-up, n=0,11 |  | -0.606 (4.1280)

7. Primary Outcome: Change From Baseline in ECG; PR Interval, QRS Duration, QT Interval and QTcF
Description: Triplicate 12-lead ECGs were obtained using an ECG machine that automatically measured PR, QRS, QT, and QT interval corrected using Fridericia's formula (QTcF) intervals. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. All participants received both treatment interventions at the same time (on different skin sites), hence data for these participants were combined.
Time Frame: Baseline (Day 1), Day 14 and follow-up (up to Day 56)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Group A-Participants With Photoprovocation Lesions | Group B-Participants With Natural Lesions
Number analyzed (Participants) | 0 | 11
Milliseconds
  PR interval, Day 14, n=0,10: number analyzed (Participants) | 0 | 10
  PR interval, Day 14, n=0,10 |  | -0.900 (5.2306)
  PR interval, Follow-up, n=0,11 |  | 3.424 (11.4174)
  QRS duration, Day 14, n=0,10: number analyzed (Participants) | 0 | 10
  QRS duration, Day 14, n=0,10 |  | -0.967 (3.4728)
  QRS duration, Follow-up, n=0,11 |  | 1.061 (3.5113)
  QT interval, Day 14, n=0,10: number analyzed (Participants) | 0 | 10
  QT interval, Day 14, n=0,10 |  | -4.467 (21.8955)
  QT interval, Follow-up, n=0,11 |  | 4.455 (17.5463)
  QTcF interval, Day 14, n=0,3: number analyzed (Participants) | 0 | 3
  QTcF interval, Day 14, n=0,3 |  | -2.739 (7.4559)
  QTcF interval, Follow-up, n=0,4: number analyzed (Participants) | 0 | 4
  QTcF interval, Follow-up, n=0,4 |  | 4.532 (10.0979)

8. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect and other situations according to medical or scientific judgement or events associated with liver injury and impaired liver function.
Time Frame: Up to Day 56
Population: Safety Population. All participants received both treatment interventions at the same time (on different skin sites), hence data for these participants were combined. Data was not collected for Group A as no participants were dosed.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A-Participants With Photoprovocation Lesions | Group B-Participants With Natural Lesions
Number analyzed (Participants) | 0 | 11
Participants
  Any AEs |  | 8
  Any SAEs |  | 1

9. Secondary Outcome: Change From Baseline in Erythema, Scaling Hyperkeratosis, Edema/Infiltration, Dyspigmentation, Modified Revised Cutaneous Lupus Erythematosus Disease Area and Severity Index (RCLASI) Activity Score and Overall RCLASI Modified Score.
Description: The score ranges for different components were; erythema [0 (absent) to 3 (dark red, purple/violaceous/crusted/hemorrhagic)], scaling/hyperkeratosis [0 (absent) to 2 (verrucous hyperkeratosis)], edema/infiltration [0 (absent) to 2 (palpable and visible)] and dyspigmentation [0 (absent) to 2 (hypo and hyper pigmentation)]. For all components, 0 (better) and 3 (worse). Modified RCLASI activity score was derived by adding score for erythema, scaling hyperkeratosis and edema/infiltration. Modified change from Baseline ranged from -7 to 7, 0 (no change), minus (better) and positive (worse). Overall RCLASI modified score was derived by summing the activity and dyspigmentation scores. Overall change from Baseline ranged from -9 to 9, 0 (no change), minus (better) and positive (worse). Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Data was not collected for Group A as no participants were dosed.
Time Frame: Baseline (Day 1), Day 14 and Day 28
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles). All participants received both treatment interventions at the same time (on different skin sites), hence data for these participants were combined.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Group A-Participants With Photoprovocation Lesions; Placebo: Participants who developed photoprovocation lesions following photoprovocation challenge were planned to be topically administered white to off-white aqueous cream of placebo. The treatments were planned to be administered at the same time on different skin sites once daily for 28 days.
- Group A-Participants With Photoprovocation Lesions; GSK2646264: Participants who developed photoprovocation lesions following photoprovocation challenge were planned to be topically administered white to off-white aqueous cream of GSK2646264 (1% weight by weight, [w/w]). The treatments were planned to be administered at the same time on different skin sites once daily for 28 days.
- Group B-Participants With Natural Lesions; Placebo: Participants with natural lesions were topically administered white to off-white aqueous cream of placebo. The treatments were administered at the same time on different skin sites once daily for 28 days.
- Group B-Participants With Natural Lesions; GSK2646264: Participants with natural lesions were topically administered white to off-white aqueous cream of GSK2646264 (1% w/w). The treatments were administered at the same time on different skin sites once daily for 28 days.
Arm/Group | Group A-Participants With Photoprovocation Lesions; Placebo | Group A-Participants With Photoprovocation Lesions; GSK2646264 | Group B-Participants With Natural Lesions; Placebo | Group B-Participants With Natural Lesions; GSK2646264
Number analyzed (Participants) | 0 | 0 | 11 | 11
Scores on a scale
  Erythema, Day 14, n=0,0,9,9: number analyzed (Participants) | 0 | 0 | 9 | 9
  Erythema, Day 14, n=0,0,9,9 |  |  | -0.8 (0.83) | -0.8 (0.83)
  Erythema, Day 28, n=0,0,10,10: number analyzed (Participants) | 0 | 0 | 10 | 10
  Erythema, Day 28, n=0,0,10,10 |  |  | -0.5 (0.71) | -0.5 (0.71)
  Scaling/Hyperkeratosis, Day 14, n=0,0,9,9: number analyzed (Participants) | 0 | 0 | 9 | 9
  Scaling/Hyperkeratosis, Day 14, n=0,0,9,9 |  |  | 0.0 (0.00) | 0.0 (0.00)
  Scaling/Hyperkeratosis, Day 28, n=0,0,10,10: number analyzed (Participants) | 0 | 0 | 10 | 10
  Scaling/Hyperkeratosis, Day 28, n=0,0,10,10 |  |  | 0.0 (0.00) | 0.0 (0.00)
  Edema/infiltration, Day 14, n=0,0,9,9: number analyzed (Participants) | 0 | 0 | 9 | 9
  Edema/infiltration, Day 14, n=0,0,9,9 |  |  | -0.2 (0.44) | -0.2 (0.44)
  Edema/infiltration, Day 28, n=0,0,10,10: number analyzed (Participants) | 0 | 0 | 10 | 10
  Edema/infiltration, Day 28, n=0,0,10,10 |  |  | -0.4 (0.52) | -0.3 (0.48)
  Dyspigmentation, Day 14, n=0,0,9,9: number analyzed (Participants) | 0 | 0 | 9 | 9
  Dyspigmentation, Day 14, n=0,0,9,9 |  |  | -0.1 (0.33) | -0.1 (0.33)
  Dyspigmentation, Day 28, n=0,0,10,10: number analyzed (Participants) | 0 | 0 | 10 | 10
  Dyspigmentation, Day 28, n=0,0,10,10 |  |  | -0.1 (0.32) | -0.1 (0.32)
  Modified RCLASI, Day 14, n=0,0,9,9: number analyzed (Participants) | 0 | 0 | 9 | 9
  Modified RCLASI, Day 14, n=0,0,9,9 |  |  | -1.0 (1.22) | -1.0 (1.12)
  Modified RCLASI, Day 28, n=0,0,10,10: number analyzed (Participants) | 0 | 0 | 10 | 10
  Modified RCLASI, Day 28, n=0,0,10,10 |  |  | -0.9 (1.20) | -0.8 (1.14)
  Overall RCLASI modified, Day 14, n=0,0,9,9: number analyzed (Participants) | 0 | 0 | 9 | 9
  Overall RCLASI modified, Day 14, n=0,0,9,9 |  |  | -1.1 (1.45) | -1.1 (1.36)
  Overall RCLASI modified, Day 28, n=0,0,10,10: number analyzed (Participants) | 0 | 0 | 10 | 10
  Overall RCLASI modified, Day 28, n=0,0,10,10 |  |  | -1.0 (1.33) | -0.9 (1.37)

10. Secondary Outcome: Maximum Observed Concentration (Cmax) of GSK2646264 in Participants With Cutaneous Lupus Erythematosus (CLE)
Description: Blood samples were collected at designated timepoints and pharmacokinetic (PK) analysis was performed. Cmax was calculated by non-compartmental analysis using WinNonlin. PK Population comprised of all participants in the safety population for whom a PK sample was obtained and analyzed.
Time Frame: Day 1 (pre-dose and 5 hours post-dose), Day 2 to Day 13, Day 14 (pre-dose), Day 21 to Day 27, Day 28 (post-dose), Day 29 to Day 42 and Follow-up (up to Day 56)
Population: PK Population. All participants received both treatment interventions at the same time (on different skin sites), hence data for these participants were combined. Data was not collected for Group A as no participants were dosed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Group A-Participants With Photoprovocation Lesions | Group B-Participants With Natural Lesions
Number analyzed (Participants) | 0 | 11
Nanogram per milliliter |  | 0.8324 (109.3)

11. Secondary Outcome: Time to Reach Maximum Observed Concentration (Tmax) of GSK2646264 in Participants With CLE
Description: Blood samples were collected at designated timepoints and PK analysis was performed. Tmax was calculated by non-compartmental analysis using WinNonlin.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | Group A-Participants With Photoprovocation Lesions | Group B-Participants With Natural Lesions
Number analyzed (Participants) | 0 | 11
Hours |  | 311.467 [4.68 to 651.92]

12. Secondary Outcome: Mean Fold Change in Messenger Ribonucleic Acid (mRNA) Expression of Interferon (IFN) Signatures in Skin Biopsies
Description: Microarray mRNA data was collected from the skin biopsy in both GSK2646264 and placebo treated lesions on Day -5 to -3 visit (Baseline) and Day 28. Fold change represents the change at Day 28 relative to Baseline for each treatment group. Analysis was conducted using mixed model with participant as a random effect and treatment as a fixed effect where treatment is set to "not applicable" at Baseline. Mean fold change and 95% confidence interval is presented for different genes and probesets. IFI16 indicated interferon, gamma-inducible protein 16, IFI44 indicated interferon-induced protein 44, IFIH1 indicated interferon induced with helicase C domain 1, IFIT1 and 3 indicated interferon-induced protein with tetratricopeptide repeats 1 and 3, MX1 indicated myxovirus (influenza virus) resistance 1, interferon-inducible protein p78 (mouse), MX2 indicated myxovirus (influenza virus) resistance 2 (mouse) and OAS indicated 2'-5'-oligoadenylate synthetase.
Time Frame: Baseline (Day -5 to -3) and Day 28
Population: Safety Population. Only those participants with data available at the specified data points were analyzed. Data was not collected for Group A as no participants were dosed.
Measure: Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Group A-Participants With Photoprovocation Lesions; Placebo | Group A-Participants With Photoprovocation Lesions; GSK2646264 | Group B-Participants With Natural Lesions; Placebo | Group B-Participants With Natural Lesions; GSK2646264
Number analyzed (Participants) | 0 | 0 | 9 | 9
Fold change
  Chemokine (C-X-C motif)Ligand10, 204533_at, Day 28 |  |  | 1.173 [-1.899 to 2.610] | -1.464 [-3.259 to 1.521]
  IFI16, 206332_s_at, Day 28 |  |  | -1.001 [-1.286 to 1.283] | -1.064 [-1.367 to 1.207]
  IFI16, 208965_s_at, Day 28 |  |  | 1.055 [-1.219 to 1.356] | -1.164 [-1.496 to 1.105]
  IFI16, 208966_x_at, Day 28 |  |  | -1.044 [-1.328 to 1.219] | -1.096 [-1.394 to 1.161]
  IFI44, 214059_at, Day 28 |  |  | 1.018 [-1.429 to 1.481] | -1.029 [-1.497 to 1.413]
  IFI44, 214453_s_at, Day 28 |  |  | 1.021 [-1.541 to 1.606] | -1.270 [-1.998 to 1.239]
  IFI44-like, 204439_at, Day 28 |  |  | 1.043 [-1.602 to 1.744] | -1.122 [-1.875 to 1.491]
  IFIH1, 1555464_at, Day 28 |  |  | 1.037 [-1.081 to 1.162] | -1.074 [-1.204 to 1.043]
  IFIH1, 216020_at, Day 28 |  |  | 1.035 [-1.062 to 1.138] | -1.044 [-1.148 to 1.053]
  IFIH1, 219209_at, Day 28 |  |  | -1.025 [-1.577 to 1.500] | -1.295 [-1.991 to 1.188]
  IFIT1, 203153_at, Day 28 |  |  | 1.011 [-1.664 to 1.701] | -1.113 [-1.872 to 1.512]
  IFIT3, 204747_at, Day 28 |  |  | 1.039 [-1.643 to 1.772] | -1.221 [-2.084 to 1.397]
  IFIT3, 229450_at, Day 28 |  |  | 1.096 [-1.457 to 1.749] | -1.138 [-1.817 to 1.402]
  Interleukin 1, alpha, 208200_at, Day 28 |  |  | 1.016 [-1.324 to 1.367] | -1.217 [-1.638 to 1.105]
  Interleukin 1, alpha, 210118_s_at, Day 28 |  |  | -1.015 [-1.117 to 1.085] | -1.169 [-1.287 to -1.062]
  Interleukin 1, beta, 205067_at, Day 28 |  |  | 1.081 [-1.145 to 1.337] | -1.131 [-1.399 to 1.094]
  Interleukin 1, beta, 39402_at, Day 28 |  |  | 1.087 [-1.166 to 1.377] | -1.094 [-1.386 to 1.158]
  Interleukin 6, 205207_at, Day 28 |  |  | 1.014 [-1.077 to 1.107] | 1.063 [-1.027 to 1.161]
  ISG15 ubiquitin-like modifier, 205483_s_at, Day 28 |  |  | -1.086 [-2.044 to 1.732] | -1.343 [-2.527 to 1.401]
  MX1, 202086_at, Day 28 |  |  | 1.059 [-1.244 to 1.395] | -1.028 [-1.354 to 1.281]
  MX2, 204994_at, Day 28 |  |  | 1.122 [-1.271 to 1.601] | -1.039 [-1.482 to 1.374]
  OAS1, 40/46 kilodalton, 202869_at, Day 28 |  |  | 1.092 [-1.219 to 1.453] | -1.168 [-1.555 to 1.139]
  OAS1, 40/46 kilodalton, 205552_s_at, Day 28 |  |  | 1.088 [-1.391 to 1.646] | -1.296 [-1.961 to 1.168]
  OAS2, 69/71 kilodalton, 204972_at, Day 28 |  |  | 1.165 [-1.347 to 1.826] | -1.157 [-1.814 to 1.355]
  OAS2, 69/71 kilodalton, 206553_at, Day 28 |  |  | 1.061 [-1.186 to 1.334] | -1.010 [-1.270 to 1.246]
  OAS2, 69/71 kilodalton, 228607_at, Day 28 |  |  | 1.065 [-1.478 to 1.676] | 1.000 [-1.574 to 1.574]
  OAS3, 100 kilodalton, 218400_at, Day 28 |  |  | 1.141 [-1.370 to 1.784] | -1.089 [-1.702 to 1.436]
  OAS3, 100 kilodalton, 232666_at, Day 28 |  |  | 1.096 [-1.274 to 1.529] | 1.109 [-1.259 to 1.548]
  OAS-like, 205660_at, Day 28 |  |  | 1.179 [-1.586 to 2.206] | -1.217 [-2.276 to 1.537]
  OAS-like, 210797_s_at, Day 28 |  |  | 1.178 [-1.508 to 2.091] | -1.112 [-1.973 to 1.597]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study treatment up to Day 56
Description: Safety Population comprised of all participants who received at least one dose of a study treatment. Data was not collected for Group A as no participants were dosed.
Arm/Group | Group A-Participants With Photoprovocation Lesions | Group B-Participants With Natural Lesions
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/11
Other Adverse Events (participants affected / at risk) | 0/0 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A-Participants With Photoprovocation Lesions (N=0) | Group B-Participants With Natural Lesions (N=11)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A-Participants With Photoprovocation Lesions (N=0) | Group B-Participants With Natural Lesions (N=11)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT02927457/SAP_000.pdf
  • Study Protocol (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT02927457/Prot_001.pdf